CLINICAL TRIAL: NCT00843544
Title: Effect of an Integrative Medicine Approach to the Management of Asthma in Adults on Quality of Life and Clinical Outcomes
Brief Title: Integrative Medicine Approach to the Management of Asthma in Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Benjamin Kligler, Beth Israel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170-05
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrative Medicine (Experimental)
  Interventions: Behavioral: Integrative Medicine
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Integrative Medicine — Participants assigned to the treatment group will begin in groups of ten. The treatment protocol will consist of six 1-2 hour sessions over a six-week period as follows:
  1. Subjects will attend a two-session class on healthy eating focused on reducing inflammation-promoting foods in the diet. All subjects will also be started on fish oil and vitamin C supplements, as well as on a supplement called Kaprex, which is an extract from hops and rosemary with anti-inflammatory action. Supplements willl be provided free of charge. Subjects will be provided with a take home supply to begin using.
  2. Subjects will attend two classes at CCHH in yoga breathing techniques and will then be provided with a CD for home study and practice
  3. Subjects will attend two guided journaling sessions at CCHH in which subjects will be asked to write for a 30-minute period about the most traumatic or stressful life experience to date.
  Arms: Integrative Medicine

SUMMARY:
The overall aim of this research project is to test the effectiveness of an integrative program, using journaling, yoga breathing instruction, and nutritional manipulation and supplementation, on quality of life and clinical outcomes in adults with asthma. An additional aim is to determine whether an integrative approach to asthma management leads to cost savings when compared to standard clinical care.Patients will be randomly assigned to either the intervention condition or a waitlist control condition. For the intervention group, all measures will be obtained at baseline, immediately after the treatment protocol is completed, and then at three month and six month intervals after the completion of the intervention. For the control group, data will be collected at the same times as the intervention group, with one exception: data collected at the completion of the treatment protocol will be replaced with data collection at six weeks post-baseline for the control group. Data will be collected using measures of quality of life (Asthma Quality of Life Questionnaire and SF-12), pulmonary function and health care utilization and expenditures.

Participants assigned to the treatment group will begin in groups of ten. The treatment protocol will consist of six 1-2 hour sessions over a six-week period as follows:

1. Subjects will attend a two-session class on healthy eating focused on reducing inflammation-promoting foods in the diet. All subjects will also be started on fish oil and vitamin C supplements, as well as on a supplement called Kaprex, which is an extract from hops and rosemary with anti-inflammatory action. Supplements willl be provided free of charge. Subjects will be provided with a take home supply to begin using.
2. Subjects will attend two classes at CCHH in yoga breathing techniques and will then be provided with a CD for home study and practice
3. Subjects will attend two guided journaling sessions at CCHH in which subjects will be asked to write for a 30-minute period about the most traumatic or stressful life experience to date.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. Class II through IV asthma sufferers will be included (mild persistent; moderate persistent; severe persistent).
3. Ability to read and write at minimum fifth grade level
4. Willing to comply with study instructions and sign an informed consent
5. English-speaking

Exclusion Criteria:

1. Pregnancy or lactation
2. Concurrent serious or life-threatening illness as determined by clinical judgment
3. Psychiatric disorder as determined by clinical judgment.
4. Inability to understand or follow the instructions associated with the clinical study as determined by clinical judgment.
5. Fish allergy or history of adverse reaction to vitamin C or fish oil as determined by clinical history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaire | Baseline, 6 weeks, 3 months, 6 months

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form-12 (SF-12) | Baseline, 6 weeks, 3 months, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Medical Center/Center for Health and Healing, New York, New York, United States

REFERENCES:
- [Derived] Kligler B, Homel P, Blank AE, Kenney J, Levenson H, Merrell W. Randomized trial of the effect of an integrative medicine approach to the management of asthma in adults on disease-related quality of life and pulmonary function. Altern Ther Health Med. 2011 Jan-Feb;17(1):10-5. PMID 21614939